CLINICAL TRIAL: NCT03005704
Title: Reversal of the Antiplatelet Effects of Ticagrelor in Combination With Aspirin, Using Normal Platelets
Acronym: REVSTARTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Paul Kruger, Dr, Hamilton Health Sciences Corporation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PopulationHRI
Record Dates: First submitted 2016-12-26; First posted 2016-12-29 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Ticagrelor; Aspirin; Platelet Dysfunction Due to Drugs; Transfusion
Keywords: Ticagrelor; Acetylsalicylic acid; Platelet transfusion; Reversal
MeSH Terms: interventions — Ticagrelor; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antiplatelet Treatment (Experimental): Subjects will be treated with five days of ticagrelor in combination with acetylsalicylic acid.
  Interventions: Drug: Antiplatelet treatment
- Control (No Intervention): Subjects will not receive antiplatelet treatment and their PRP will be used as the source of untreated platelets in laboratory mixing studies.

INTERVENTIONS:
Drug: Antiplatelet treatment — Subjects will be treated with ticagrelor in combination with acetylsalicylic acid for five days. Ticagrelor will be administered at a loading dose of 180 mg, followed by 90 mg twice daily maintenance dose. Acetylsalicylic acid will be administered at a dose of 81 mg daily.
  Other Names: Ticagrelor and acetylsalicylic acid
  Arms: Antiplatelet Treatment

SUMMARY:
The specific objective of this study is to investigate the potential for normal platelets to reverse the inhibition of platelet aggregation in patients treated with ticagrelor in combination with aspirin.

DETAILED DESCRIPTION:
Ticagrelor is one of three commercially available antiplatelet adenosine diphosphate (ADP) antagonists (the other two are clopidogrel and prasugrel). They exert their antiplatelet effects by binding to P2Y12 receptors on the platelet surface. Ticagrelor is used in combination with aspirin to prevent and treat thrombosis in patients with acute coronary syndrome, particularly after stent implantation. ADP antagonists are combined with aspirin because aspirin blocks platelet aggregation by preventing thromboxane production, and blocking two different pathways leads to greater efficacy than either drug used alone. Recent clinical trials indicate ticagrelor in combination with aspirin is more effective for prevention of thrombotic events in patients with symptomatic coronary artery disease than aspirin in combination with clopidogrel, but causes significantly more bleeding. The improved efficacy and reduced safety occurs because ticagrelor causes greater inhibition of ADP-mediated platelet activation. The latter can be reliably measured in the laboratory.

Management of patients who bleed while taking an ADP antagonist in combination with aspirin is challenging because there is no specific antidote, Platelet transfusion has the potential to reverse the effects of clopidogrel or prasugrel and aspirin, but these findings cannot be extrapolated to ticagrelor in combination with aspirin because the pharmacokinetic and pharmacodynamic effects of ticagrelor differ.

Aspirin, clopidogrel active metabolite, and prasugrel active metabolite have half-lives of 15-20 minutes, 30 minutes, and four hours respectively. They are irreversible platelet inhibitors which bind to and permanently block platelet function. After their drug elimination, new platelets which enter the circulation from megakaryocytes in the bone marrow are unaffected. Therefore, after elimination, newly transfused platelets have the potential to restore haemostasis. In contrast, ticagrelor, a reversible platelet inhibitor, has a longer half-life (7.7 to 14.1 hours). As a result of its longer half-life, newly added platelets (both from the bone marrow and transfused platelets) are inhibited by ticagrelor for at least 24 hours after the last dose. Therefore, reversing platelet inhibition and controlling excessive bleeding associated with ticagrelor by platelet transfusion poses a greater challenge than with clopidogrel and prasugrel. Nevertheless, because of its greater efficacy, ticagrelor is preferred over clopidogrel in high risk patients.

Previous studies of platelet transfusion and ev vivo mixing within 24 hours of drug administration have shown than the inhibition of ADP-mediated platelet activation by clopidogrel and prasugrel, but not ticagrelor can be reversed or modulated by the addition of donor platelets. Although reversing the platelet inhibitory effects of ticagrelor might not be possible within 24 hours of stopping the drug, it should be possible in the days that follow. This has not been examined. Accordingly, we propose to perform a study in which we systematically evaluate inhibition of ADP mediated platelet activation, a reliable measure of ticagrelor's antiplatelet activity, when donor platelets are added to the platelets of subjects treated with ticagrelor at time intervals up to 96 hours after their last dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* At least 18 years of age
* No history of cardiovascular disease
* Not taking antiplatelet therapy prior to participation

Exclusion Criteria:

* Known thrombocytopenia, other coagulation disorder such as von Willebrand's disease, haemophilia
* Allergy or intolerance to ticagrelor or aspirin (if known)
* Consumption of drugs within the preceding fourteen days that potentially can interfere with metabolism of ticagrelor through CYP3A4, CYP3A or P-glycoprotein (eg, ketoconazole, clarithromycin, nefazodone, ritonavir, atazanavir, diltiazem, amprenavir, aprepitant, erythromycin, fluconazole, verapamil, rifampicin, dexamethasone, phenytoin, carbamazepine, phenobarbital, cyclosporine, simvastatin, atorvastatin, tolbutamide, digoxin)21
* Previous transfusion or pregnancy (because of potential alloimmunisation)
* Pregnant or trying to conceive, or breastfeeding
* Unable or unwilling to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Reversal of platelet inhibition | 5 days
  The primary outcome is to measure the efficacy of untreated platelets in reversing the platelet inhibition due to ticagrelor in combination with aspirin by ex vivo mixing studies. Increase in platelet aggregation will be measured by light transmission aggregometry after stimulation by adenosine diphosphate, arachidonic acid, and collagen.

SECONDARY OUTCOMES:
Timing of reversal of platelet inhibition | 5 days
  The secondary outcome measure is to determine the time point post cessation at which untreated donor platelets reverse the antiplatelet effect of ticagrelor in combination with aspirin.

CONTACTS AND LOCATIONS:
Locations (1):
- Population Health Research Institute, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No